CLINICAL TRIAL: NCT02767479
Title: Comparison of Rabeprazole and Esomperazole for the Eradication of H. Pylori (CREATION Study)
Brief Title: Comparison of Rabeprazole and Esomperazole for the Eradication of H. Pylori
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamamatsu University (Other)
Responsible Party: Principal Investigator, Takahisa Furuta, Professor, Hamamatsu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-125
Record Dates: First submitted 2014-12-10; First posted 2016-05-10 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: H. Pylori Infection
Keywords: eradication rates; rabeprazole; esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rabeprazole group (Active Comparator): rabeprazole-based regimen. This group is treated with rabeprazole 10 mg bid, AMPC 750 mg bid and CAM 200 mg bid for 1 week. Success or Failure of eradication of H. pylori is assessed by 13C-UBT 1 month after the treatment.
  Interventions: Drug: rabeprazole-based regimen
- esomeprazole group (Active Comparator): 'esomeprazole^based regimen. This group is treated with esomeprazole 20 mg bid , AMPC 750 mg bid and CAM 200 mg bid for 1 week. Success or Failure of eradication of H. pylori is assessed by 13C-UBT 1 month after the treatment.
  Interventions: Drug: esomeprazole^based regimen

INTERVENTIONS:
Drug: rabeprazole-based regimen — This group is treated with rabeprazole 10 mg bid, AMPC 750 mg bid and CAM 200 mg bid for 1 week. Success or Failure of eradication of H. pylori is assessed by 13C-UBT 1 month after the treatment.
  Other Names: RAC
  Arms: rabeprazole group
Drug: esomeprazole^based regimen — This group is treated with esomeprazole 20 mg bid , AMPC 750 mg bid and CAM 200 mg bid for 1 week. Success or Failure of eradication of H. pylori is assessed by 13C-UBT 1 month after the treatment.
  Other Names: EAC
  Arms: esomeprazole group

SUMMARY:
Patients infected with H. pylori are treated with rabeprazole 10 mg bid, AMPC 750 mg bid and CAM 200 mg bid or esomeprazole 20 mg bid, AMPC 750 mg bid and CAM 200 mg bid. Eradication rates are compared. Patients who have ever failed in eradication by CAM-based regimen are treated with rabeprazole 10 mg bid, AMPC 750 mg bid and MNZ 250 mg bid or esomeprazole 20 mg bid, AMPC 750 mg bid and MNZ 250 mg bid.

DETAILED DESCRIPTION:
Patients infected with H. pylori are treated with rabeprazole 10 mg bid, AMPC 750 mg bid and CAM 200 mg bid or esomeprazole 20 mg bid, AMPC 750 mg bid and CAM 200 mg bid. Eradication rates are compared. Patients who have ever failed in eradication by CAM-based regimen are treated with rabeprazole 10 mg bid, AMPC 750 mg bid and MNZ 250 mg bid or esomeprazole 20 mg bid, AMPC 750 mg bid and MNZ 250 mg bid. CYP2C19 genotypes and susceptibility to CAM are genetically measured. Other factors are also analyzed with reference to eradication rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with H. pylori who can undergo the eradication therapy

Exclusion Criteria:

* Patients with severe other disorders, cannot undergo eradication therapy, refuses to participate to the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Eradication rates of H. pylori | At 4 weeks after treatment
  Success or failure eradication of H. pylori was judged based on the 13C-urea breath test performed 1 month after the treatment.
influence of CYP2C19 genotypes on the eradication rates of H. pylori | At 4 weeks after treatment
  influence of CYP2C19 genotypes on the eradication rates of H. pylori are analyzed. CYP2C19 genotypes are classified to the three groups, rapid metabolizer (RM), intermiediate metabolizer (IM) and Poor metabolizer (PM). Because esomperazole is metabolized by CYP2C19, the effects of esomeprazole is influenced by genotypes of CYP2C19. The eradication rates in RMs, IMs and PMs are compared.
Influences of susceptibility of H. pylori strains to clarithromycin (CAM) on the eradication rates of H. pylori | At 4 weeks after treatment
  Influences of susceptibility to clarithromycin on eradication rates of H. pylori are analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan